CLINICAL TRIAL: NCT01875653
Title: Phase III, Randomized, Double-Blind, Multicenter Trial of Autologous Dendritic Cells and Irradiated Autologous Tumor Cells In Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) vs. Autologous Peripheral Blood Mononuclear Cells (PBMCs) In GM-CSF for The Treatment Of Metastatic Melanoma
Brief Title: Autologous Dendritic Cell-Tumor Cell Immunotherapy for Metastatic Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-CA-P01; 2015-001984-38 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-12 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Stage IV Melanoma; Stage III Melanoma
Keywords: metastatic melanoma; dendritic cells; immunotherapy; Granulocyte-Macrophage Colony Stimulating Factor; overall survival; autologous; peripheral blood mononuclear cells; treatment; phase 3; tumor cells
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous PBMCs in GM-CSF (MC) (Active Comparator): DOSE/ROUTE/REGIMEN:
  1. Treatment Duration: Doses of MC will be administered subcutaneously weekly for 3 consecutive weeks, then monthly for the next 5 months.
  2. Dosage: Each dose of MC contains approximately 10 million cells. Each dose is suspended in 500 mcg GM-CSF prior to administration.
  3. Mode of Administration: Subcutaneous (SC) injections.
  Interventions: Biological: Autologous PBMCs in GM-CSF (MC)
- Autologous Dendritic Cell-Tumor Cell Immunotherapy (DC-TC) (Experimental): DOSE/ROUTE/REGIMEN:
  1. Treatment Duration: Doses of DC-TC will be administered subcutaneously weekly for 3 consecutive weeks, then monthly for the next 5 months.
  2. Dosage: Each dose of DC-TC contains approximately 10-20 million cells. Each dose is suspended in 500 mcg GM-CSF prior to administration.
  3. Mode of Administration: Subcutaneous (SC) injections.
  Interventions: Biological: Autologous Dendritic Cell-Tumor Cell Immunotherapy (DC-TC)

INTERVENTIONS:
Biological: Autologous Dendritic Cell-Tumor Cell Immunotherapy (DC-TC) — Comparison of a cancer treatment containing patient specific irradiated tumor cells mixed with antigen presenting immune cells suspended in an immune system stimulant vs. a cancer treatment containing patient specific immune cells suspended in an immune system stimulant
  Other Names: DC-TC; MAC-VAC; Autologous Dendritic Cells Loaded With Irradiated Autologous Tumor Cells In GM-CSF; Melapuldencel-T
  Arms: Autologous Dendritic Cell-Tumor Cell Immunotherapy (DC-TC)
Biological: Autologous PBMCs in GM-CSF (MC) — Comparison of a cancer treatment containing patient specific irradiated tumor cells mixed with antigen presenting immune cells suspended in an immune system stimulant vs. a cancer treatment containing patient specific immune cells suspended in an immune system stimulant
  Arms: Autologous PBMCs in GM-CSF (MC)

SUMMARY:
The purpose of this research is to evaluate the safety and effectiveness of tumor cell therapy.

This research study is evaluating if a patient-specific experimental therapy for metastatic melanoma will lengthen survival with minimal harmful effects. It is called an experimental therapy (or "study therapy") because it is not yet approved by the U.S. Food and Drug Administration (FDA). This research study will use the patient's own tumor cells,the patient's own dendritic cells (a type of immune cell), and a granulocyte-macrophage colony stimulating factor (GM-CSF, a type of growth factor). GM-CSF is a natural growth factor that stimulates growth of white blood cells in the body. Since 1991, GM-CSF has been used as a standard treatment to help increase the number of white blood cells after chemotherapy.

The patient's dendritic cells are grown in a test-tube with the patient's tumor cells and the growth factor. The resulting solution is called the study therapy. The intent of the study therapy is to make the dendritic cells more effective at fighting the tumor when they are injected back into the patient.

DETAILED DESCRIPTION:
Learn more about this clinical trial at http://TheIntusStudy.com. Type or copy and paste http://TheIntusStudy.com in your browser window.

ELIGIBILITY:
INCLUSION CRITERIA:

Pre-Treatment Phase: Tissue Procurement and Establishment of Tumor Cell Line

1. Histologic diagnosis of invasive melanoma.
2. Measurable metastatic melanoma with at least one lesion amenable to -resection Stage III: recurrent regional disease, including regional disease with no known primary.

   Stage IV: distant metastatic melanoma.
3. Age 18 years and older.
4. Sign the "Tissue Consent", the pre-Clinical Informed Consent for Melanoma Tissue Procurement and initiation of cell line effort granting Caladrius permission to cryopreserve the tumor and/or to initiate an autologous tumor cell line from excess tissue that has been removed during a medical procedure (e.g., surgically excised).
5. Initiation of Autologous Tumor Cell Line. Caladrius must have received a viable melanoma tumor tissue specimen that has been obtained and processed according to company SOPs to ensure tissue viability. The cell line can be initiated with either a specimen of fresh tumor or tumor that has been previously cryopreserved.

Treatment Phase

1. Successful establishment of an autologous melanoma cell line by Caladrius.
2. Patients with multiple depots of distant metastatic disease must have previously received at least one or more of the following standard treatments: interleukin 2 (IL-2), or ipilimumab, or vemurafenib (if tumor expresses the V600E mutation), or dacarbazine or temozolomide, if not mutated for the V600E mutation, and not felt to be medically appropriate for IL-2 or ipilimumab. These may have been given alone, or in combination with other agents.
3. Medical fitness to undergo a leukapheresis, including peripheral venous access or access by central vein if necessary.
4. Medical fitness for participation in a phase III clinical trial.

   * a. ECOG performance status of 0 or 1.
   * b. Adequate bone marrow function: absolute neutrophil count (ANC) greater than 1000/mm (3), hematocrit greater than 30%, platelet count greater than 100,000/mm (3), no ongoing transfusion requirements.
   * c. Adequate hepatic function: total bilirubin less than 2.0 mg/dL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 3 times the upper limit of normal (ULN), albumin greater than 3 g/dL.
   * d. Adequate kidney function: creatinine less than or equal to 2.0 mg/dL.
   * e. Negative pregnancy test for woman of childbearing potential and use of effective contraception (hormonal or barrier method of birth control) during therapy (women of childbearing potential and men).
5. Extent of disease established within 4 weeks of randomization.

   * a. History and Physical Exam by a licensed practitioner.
   * b. Fludeoxyglucose(FDG)-based PET/CT or PET scan and CT scan.
   * c. Brain MRI demonstrating no new untreated or uncontrolled metastases.
6. Recovery from previous therapies.

   * a. At least four weeks (28 days) must have elapsed since any prior systemic therapy at the time of the first dose (six weeks for anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4), and any toxicities experienced must have recovered to a grade 1 or less (except for alopecia or vitiligo).
   * b. More than three weeks (at least 22 days) since radiation therapy at the time of the first dose (7 days for single-dose stereotactic radiotherapy such as gamma knife) and recovery from acute toxicities. Patients treated with whole brain radiation must wait at least 22 days after completion of radiation and have radiographic confirmation of lack of progression before proceeding to randomization.

EXCLUSION CRITERIA:

Pre-Treatment Phase: Tissue Procurement and Establishment of Tumor Cell Line

1. Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
2. Lack of a metastatic melanoma lesion that can be resected.

Treatment Phase

1. Known positive for hepatitis B or C or HIV.
2. Pregnant or lactating women.
3. Underlying cardiac disease associated with known myocardial dysfunction, or active treatment with digoxin or other medications being given to treat heart failure, or unstable angina related to atherosclerotic cardiovascular disease.
4. Diagnosis of any other invasive cancer that requires ongoing treatment or for which there is evidence of active disease.
5. Active, unresolved infection and/or receiving concurrent treatment with parenteral antibiotics (patients are eligible after antibiotics have been discontinued for at least 7 days prior to first dose and evidence of infection has resolved).
6. Other active medical condition that could be imminently life threatening, in the opinion of the investigator, including no active blood clotting or bleeding diathesis.
7. New or uncontrolled brain metastases or leptomeningeal disease and/or taking pharmacological doses of corticosteroids. Brain metastases treated by gamma knife or stereotactic radiotherapy are considered controlled, unless patient requires pharmacologic doses of corticosteroids. It is recognized that tumor necrosis may be confused with tumor progression in interpretation of Brain MRI.
8. Known autoimmune disease, immunodeficiency, or disease process that involves the use of immunosuppressive therapy.
9. Taking other anticancer therapy.
10. Received another investigational drug within 28 days of the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 52 months
  The time frames are estimated time in months (rounded up to the nearest month) from the start of study. The time estimates for the analyses are based on enrolling approximately 250 patients over a 34.8 months period and having a follow up of approximately 17 months after the last patient is enrolled.

SECONDARY OUTCOMES:
Adverse Events as a Measure of Safety and Tolerability | 52 months
  * Adverse Events monitoring to assess safety and tolerability
  * History & physical examination, vital signs, clinical laboratory tests (safety), and other tests as clinically indicated adverse event monitoring to assess safety and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Caladrius Biosciences
Locations (17):
- United States (17):
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - Newport Beach, California
  - Orange, California
  - Santa Monica, California
  - Aurora, Colorado
  - Goshen, Indiana
  - Louisville, Kentucky
  - Marrero, Louisiana
  - Baltimore, Maryland
  - Hackensack, New Jersey
  - Cincinnati, Ohio
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Dallas, Texas

REFERENCES:
- [Derived] Javed A, Sato S, Sato T. Autologous melanoma cell vaccine using monocyte-derived dendritic cells (NBS20/eltrapuldencel-T). Future Oncol. 2016 Mar;12(6):751-62. doi: 10.2217/fon.16.13. Epub 2016 Feb 3. PMID 26837440